CLINICAL TRIAL: NCT07342023
Title: Contribution of GFAP and UCH-L1 Assays in Whole Blood to Optimizing Personalized Care for "Repeated Fallers" Hospitalized in Geriatric Wards
Acronym: BACHUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CH Riom (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2025 SAPIN (BACHUS); 2025-A02166-43 (Other: 2025-A02166-43)
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fallers Aged 60 Years and Older; Biomarkers / Blood; Intracranial Bleeding
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm (Experimental): The BACHUS study, a prospective single-center study, focuses on a population of patients aged 75 years and older who are hospitalized after recurrent falls. The objective is to evaluate the performance of an innovative, personalized biological screening strategy to detect intracranial hemorrhages, as an alternative to brain CT scanning, which is often difficult to access within the required time frame in elderly patients. Patients included in the study will undergo two blood measurements of the biomarkers GFAP and UCH-L1, performed on whole blood using a portable device such as the i-Stat Alinity.
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — Patients included in the study will undergo two blood measurements of the biomarkers GFAP and UCH-L1 performed on whole blood using a portable device such as the i-Stat Alinity®. The first measurement will be performed within 72 hours of admission to establish an individual baseline value. After a fall with confirmed or suspected head trauma, when a brain CT scan is deemed necessary by the referring physician, a new measurement of GFAP and UCH-L1 biomarkers will be performed on whole blood, preferably before transfer to the CT scanner, ideally between 6 and 12 hours after the fall according to HAS recommendations, followed by the brain CT scan to detect any intracranial bleeding.

SUMMARY:
The BACHUS study focuses on a population of patients aged 75 years and older who are hospitalized after recurrent falls. The objective is to evaluate the performance of an innovative, personalized biological screening strategy to detect intracranial hemorrhages, as an alternative to brain CT scanning, which is often difficult to access within the required time frame in elderly patients.

Patients included in the study will undergo two blood measurements of the biomarkers GFAP and UCH-L1 performed on whole blood using a portable device such as the i-Stat Alinity. The first measurement will be performed within 72 hours of admission in order to establish an individual baseline value, given the impossibility of relying on average reference values in this population, which is subject to variability in biomarker levels due to confounding factors.

In the event of a new fall during hospitalization, and when a brain CT scan is deemed necessary by the referring physician, a second measurement will be performed within the time window recommended by the French National Authority for Health (HAS) (6 to 12 hours after the fall), ideally before the CT scan. Apart from the addition of this blood sample, the study will not modify usual patient management, with the decision to perform a CT scan remaining at the clinician's discretion.

The primary endpoint is the diagnostic performance of this personalized strategy (sensitivity, specificity, predictive values) compared with brain CT scanning, which remains the reference standard. The results will make it possible to estimate the number of CT scans that could be avoided. Secondary endpoints will allow further refinement of the analysis according to patient profile (age, sex, cognitive status, anticoagulant therapy, nutritional status, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged 75 years and older, cared for in the short-stay geriatric unit at Guy Thomas Hospital in Riom
* Recurrent fallers (more than one fall per week)
* Informed consent from the patient or their designated representative for patients unable to write but capable of understanding and consenting to participate in the study
* Enrollment in a Social Security health insurance scheme

Exclusion Criteria:

* Fall occurring before the reference biomarker measurement
* Presence of an intracranial hemorrhage confirmed by CT scan at admission
* Ischemic or hemorrhagic stroke
* Inability to perform the two blood samples required by the protocol due to very limited venous access
* End-of-life situation
* Adults under legal protection (guardianship, curatorship, deprivation of liberty, or judicial protection)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Determination of the specificity, sensitivity, positive predictive value, and negative predictive value of the personalized biological strategy | From enrollment until the end of hospitalization, for a maximum duration of 28 days
  Establishment of the clinical performance of a personalized biological strategy based on the combined measurement of the biomarkers GFAP and UCH-L1 in whole blood for the detection of intracranial hemorrhages in hospitalized patients aged 75 years and older with recurrent falls.

SECONDARY OUTCOMES:
Clinical performance according to patient characteristics: stratification | From enrollment until the end of hospitalization, for a maximum duration of 28 days.
  Determination of the clinical performance of the personalized biological strategy according to the following criteria: sex, age group (75-85 years; 85-95 years; over 95 years), cognitive impairment, presence of anticoagulant therapy, nutritional status, renal impairment, fall-risk profile, or characteristics of intracranial hemorrhages.
Analysis of the organizational impact | From enrollment until the end of hospitalization, for a maximum duration of 28 days
  Estimation of the number of negative brain CT scans that could be avoided using the personalized biological strategy, compared with the conventional CT-based strategy

CONTACTS AND LOCATIONS:
Overall Officials: Clément Lahaye, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- Ch de Riom, Riom, France

IPD SHARING:
Plan to Share IPD: Undecided